CLINICAL TRIAL: NCT02044861
Title: Phase 1 Open-Label, Dose Escalation, Multi-Center Study of ACT-PFK-158, 2HCl in Patients With Advanced Solid Malignancies
Brief Title: Phase 1 Safety Study of ACT-PFK-158, 2HCl in Patients With Advanced Solid Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Advanced Cancer Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT-PFK-01
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — PFK158

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACT-PFK-158 (Experimental): dose escalation
  Interventions: Drug: PFK-158

INTERVENTIONS:
Drug: PFK-158 — IV dose escalation

SUMMARY:
ACT-PFK-158 is a novel anti-cancer agent that inhibits glucose uptake in cancer cells. The primary objective of the study will be to determine the maximum tolerated dose (MTD) and to describe any dose limiting toxicity. The secondary objectives of the study will be to determine the safety profile of the drug, to determine the pharmacokinetic profile, to identify any anti-tumor activity, and to determine the pharmacodynamic profile of ACT-PFK-158.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological evidence of solid malignancy.
2. Patients must have:

   * a. Have advanced solid tumors that are refractory to established therapies known to provide clinical benefit for the malignancy in question, OR
   * b. Be intolerant of established therapies known to provide clinical benefit for the malignancy in question
3. Patients enrolled in the dose-expansion part of the trial must have at least one lesion that may qualify as a target lesion based on the RECIST 1.1 criteria.
4. Patient is ambulatory with an ECOG performance status of 0, 1 or 2 and an estimated life expectancy of > 3 months.
5. Patient is 18 years and older.
6. Patients or their legal representatives must have the ability to read, understand and provide written informed consent for the initiation of any study related procedures.
7. Patients must have adequate bone marrow reserve as evidenced by:

   * a. WBC > 3,000/µL
   * b. Absolute neutrophil count (ANC) ≥ 1,500/µL
   * c. Platelet count ≥ 100,000/µL
   * d. Hemoglobin ≥ 9 gm/dL.
8. Patients must have adequate renal function as evidenced by a serum creatinine ≤ 1.5 X ULN for the reference laboratory OR a calculated creatinine clearance of ≥ 60 mL/min by the Cockroft-Gault equation.
9. Patients must have adequate hepatic function as evidenced by AST and ALT values ≤ 3 X ULN (≤ 5 X ULN if the liver is known to be involved by metastatic disease) and serum total bilirubin values of ≤ 1.5 X ULN for the reference laboratory.
10. Patients must have INR and PTT values ≤ 1.5X ULN for the reference laboratory.
11. Patients must be recovered from the effects of any prior chemotherapy, radiotherapy or surgery (i.e., toxicity no worse than Grade 1); for patients who have been on monoclonal antibody therapy, at least one half-life or 4 weeks (whichever is shorter) should have elapsed prior to the first scheduled day of dosing with PFK-158.
12. Patients on prior investigational agents must wait at least 5 half-lives before enrollment into the trial, or 4 weeks if the half-life of the investigational agent is not known.
13. Female patients of childbearing potential must have a negative pregnancy test within 7 days of the start of treatment.
14. Women of childbearing potential and men with female sexual partners of childbearing potential must agree to use an effective method of contraception (e.g., oral contraceptives, double-barrier methods such as a condom and a diaphragm, intrauterine device) during the study and for 90 days following the last dose of study medication or to abstain from sexual intercourse for this time; a woman not of childbearing potential is one who has undergone bilateral oophorectomies or who is post-menopausal, defined as no menstrual periods for 12 consecutive months.

Exclusion Criteria:

1. Patients with an active infection or with a fever ≥ 38.5°C within 3 days of the first scheduled day of dosing.
2. Patients with primary CNS tumors as well as patients with CNS metastases are excluded.
3. Patients with known hypersensitivity to any of the components of PFK-158.
4. Patients who are receiving investigational therapies or who have been treated with investigational therapies or investigational devices within 5 half-lives of the investigational therapy or 4 weeks of first scheduled day of dosing with PFK-158 if the half-live of the investigational agent is not known.
5. Uncontrolled hypertension as defined by SBP > 160 mm/Hg or DBP > 100 mm/Hg despite medical therapy.
6. Subjects with diabetes.
7. Patients who require pharmacologic doses of corticosteroids; replacement, topical, ophthalmologic and inhalational steroids are permitted.
8. Patients who require coumadin administration.
9. Patients with mean QTcF values of > 470 msec (in females) or > 450 msec (in males) following 3 ECGs conducted 5 minutes apart from each other; patients who are known to have congenital prolonged QT syndromes; or patients who are on medications known to cause prolonged QT intervals on ECG.
10. Patients with clinically significant cardiovascular co-morbidities including: congestive heart failure (New York Heart Association class III-IV heart disease), unstable angina pectoris, cardiac arrhythmias requiring medication or a pacemaker; myocardial infarction within the past six months; stroke within the past 6 months; or hypertension requiring more than 2 medications for blood pressure control.
11. Patients with any other concurrent uncontrolled illness, including mental illness or substance abuse, which may interfere with the ability of the patient to cooperate and participate in the trial; other examples of such conditions would include COPD or diabetes mellitus that has required 2 or more hospitalizations in the last year; severe peripheral vascular disease; poorly controlled auto-immune conditions; recent serious trauma.
12. Grade 2 or higher peripheral neuropathy.
13. Patients currently known to be positive for, HIV, hepatitis B or C.
14. Patients who are pregnant or lactating.
15. Concurrent or recent (within 1 month) use of thrombolytic agents, or full-dose anticoagulants (except to maintain patency of preexisting, permanent indwelling IV catheters). Of note, therapy with low-molecular weight heparin is acceptable as long as the INR < 2.0.
16. Significant traumatic injury within the past 4 weeks.
17. Patients who are in-patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | End of cycle 1 (an average of 1 month)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Lombardi Comprehensive Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - MD Anderson Cancer Center, Houston, Texas
  - UT Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Aden D, Sureka N, Zaheer S, Chaurasia JK, Zaheer S. Metabolic Reprogramming in Cancer: Implications for Immunosuppressive Microenvironment. Immunology. 2025 Jan;174(1):30-72. doi: 10.1111/imm.13871. Epub 2024 Oct 27. PMID 39462179